CLINICAL TRIAL: NCT03451305
Title: Postrual Reduction With Pillow in Osteoporotic Vertebral Fractures: a Randomized, Prospective Study
Brief Title: Postrual Reduction With Pillow in Osteoporotic Vertebral Fracture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Principal Investigator, vghtpe user, Department of orthopedics, Taipei Veterans General Hospital, Taiwan
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 2017-05-005C
Record Dates: First submitted 2018-02-07; First posted 2018-03-01 (Actual); Last update posted 2018-03-01 (Actual); Status verified 2018-02

CONDITIONS: Compression Fracture Spine; Osteoporosis Fracture
Keywords: Compression fracture, postural reduction, vertebroplasty
MeSH Terms: conditions — Osteoporotic Fractures; Fractures, Compression

STUDY DESIGN:
Intervention Model Description: Patients with single level osteoporotic compression fracture
Who Masked: Investigator
Masking Description: Patients eligible for the study were selected by an independent research assistant. The study was explained, and informed consent was obtained from patients before the surgery. Using a randomization sequence, the patients were assigned to the international or control group. The attending surgeons and patients were blinded before the surgery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pillow group (Experimental): Before surgery, with the patient lying in the supine position, a soft pillow was placed under the segment of the collapsed vertebrae, which resulted in a hyperextension position. 12 hours duration suggested from 11:00 pm 1 night before the surgery till next day.
  Interventions: Other: Pillow
- No pillow group (No Intervention): No intervention was given in this group before surgery.

INTERVENTIONS:
Other: Pillow — A soft pillow was placed under the segment of the collapsed vertebrae, which resulted in a hyperextension position
  Arms: Pillow group

SUMMARY:
Vertebroplasty in the symptomatic osteoporotic vertebral fracture has become increasingly popular. However, there have been some limitations in restoring the height of the collapsed vertebrae and in preventing the leaking of cement. In the severely collapsed vertebrae of more than two thirds of their original height, vertebroplasty is regarded as a contraindication. We tried postural reduction using a soft pillow under the compressed level. This study was undertaken to investigate the effectiveness of the combination of postural reduction and vertebroplasty for re-expansion and stabilization of the osteoporotic vertebral fractures. single level vertebral compression fracture were treated with postural reduction followed by vertebroplasty. We analyzed the degree of re-expansion according to the onset duration.

ELIGIBILITY:
Inclusion Criteria:

* Single level osteoporotic compression fracture of thoracic and lumbar spine

Exclusion Criteria:

* Can't tolerate the postural reduction by pillow
* Pathological spine fracture caused by tumor, infection.
* Multiple spine fractures
* Patient presented with neurological. deficits

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-01-23 (Actual); Primary Completion 2019-05-23 (Estimated); Study Completion 2019-05-23 (Estimated)

PRIMARY OUTCOMES:
Sagittal plane contour | 6 months of post-operative follow up
  Sagittal plane measurement by measuring the Cobb angle of the injured vertebral on lateral radio-graphs

SECONDARY OUTCOMES:
Functional outcome | 6 months of post-operative follow up
  Visual Analogue Scale This is a pain scale, 10 scoes is the worest pain ever. 0 scores is no pain

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan

REFERENCES:
- [Background] Rao RD, Singrakhia MD. Painful osteoporotic vertebral fracture. Pathogenesis, evaluation, and roles of vertebroplasty and kyphoplasty in its management. J Bone Joint Surg Am. 2003 Oct;85(10):2010-22. No abstract available. PMID 14563813
- [Background] Lee JH, Lee DO, Lee JH, Lee HS. Comparison of radiological and clinical results of balloon kyphoplasty according to anterior height loss in the osteoporotic vertebral fracture. Spine J. 2014 Oct 1;14(10):2281-9. doi: 10.1016/j.spinee.2014.01.028. Epub 2014 Jan 23. PMID 24462536
- [Result] Chin DK, Kim YS, Cho YE, Shin JJ. Efficacy of postural reduction in osteoporotic vertebral compression fractures followed by percutaneous vertebroplasty. Neurosurgery. 2006 Apr;58(4):695-700; discussion 695-700. doi: 10.1227/01.NEU.0000204313.36531.79. PMID 16575333